CLINICAL TRIAL: NCT06823544
Title: A Comparative Single Blind Clinical Study on the Effect of Alvogyl, Eugenol, and Nigella Sativa (Black Seed Oil) for Alveolar Osteitis.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Bilal, Principal Investigator, HITEC-Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bilalkhan321@gmail.com
Record Dates: First submitted 2025-01-19; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Alveolar Osteitis
Keywords: Alveolar Osteitis; Alvogyl; Black seed oil; Eugenol; Extraction socket
MeSH Terms: conditions — Dry Socket | interventions — butyl aminobenzoate, eugenol, iodoform, spearmint oil drug combinations; Eugenol; Nigella sativa oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Alvogyl (Experimental): this group will be assigned Alvogyl as treatment drug
  Interventions: Drug: Alvogyl
- Eugenol (Experimental): this group will be assigned Eugenol as treatment drug
  Interventions: Drug: Eugenol
- Black Seed Oil (Experimental): this group will be assigned Nigella Sativa as treatment drug
  Interventions: Drug: Nigella Sativa Oil

INTERVENTIONS:
Drug: Alvogyl — this is standard treatment drug
  Arms: Alvogyl
Drug: Eugenol — this not standard drug for the treatment of Alveolar Osteitis but an antiseptic agent
  Arms: Eugenol
Drug: Nigella Sativa Oil — it not standard medicine for Alveolar Osteitis. it is a herbal medicine
  Arms: Black Seed Oil

SUMMARY:
Dry socket the unscientific term also known as alveolar or fibrinolytic osteitis is the most common postoperative complication following tooth extraction.

Treatment of Alveolar osteitis can be either pharmacological on non-pharmacological. Management can be by irrigation, surgical intervention and placement of medicated dressing such as topical anti-bacterial, topical anesthetics and obtundants or combination of these three.this study aims to find the best and effective treatment for dry socket comparing Alveogyl, Eugenol and Black seed oil at this institution.

DETAILED DESCRIPTION:
Dry socket the unscientific term also known as alveolar or fibrinolytic osteitis is the most common postoperative complication following tooth extraction. Dry socket lesion occur in approximately 1% to 5% of all extraction and up to 38% of mandibular third molar extractions. The etiology of dry socket is not yet fully understood, however the disintegration of the blood clot at the site of the tooth extraction fails to develop i.e. fibrinolysis is widely accepted as the primary mechanism or it dislodges before wound has healed. Various factors have been associated with an increase of dry socket, although some of them remain controversial and many include difficult or traumatic extractions, oral hygiene, smoking, Gender (female), extraction site, previous dry socket history, while incidence can be reduced with the chlorhexidine rinse and gel of alveolar osteitis.

Treatment of Alveolar osteitis can be either pharmacological on non-pharmacological. Management can be by irrigation, surgical intervention and placement of medicated dressing such as topical anti-bacterial, topical anesthetics and obtundants or combination of these three. Out of these Alveogyl is the still the material of choice in terms of pain relief, wound healing and low incidence of dry socket as compared to honey, zinc oxide eugenol and cutanplast , however in some recent studies a mixture of Nigella sativa powder and oil showed that it is more efficacious dressing material for the management of dry socket compared to alvogyl, it provided immediate and complete pain relief and fewer number of repeated visits needed while in some neocane was the most suitable dressing material for the management of dry socket by virtue of shorter time required for the complete pain relief, fewer visits required and faster clinical healing. Based on the previous data, we decided to conduct a study to evaluate the effectiveness of nigella sativa (black seed oil) for the treatment of dry socket compared to alveogyl and eugenol both. To the best of our knowledge, this is the first comparative study of nigella sativa oil for the treatment of dry socket at Oral and maxillofacial surgery department, HITEC dental college, Taxila and is aimed to find the best and effective treatment for dry socket comparing Alveogyl, Eugenol and Black seed oil at this institution.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 16, from both genders, who had their teeth extracted and were clinically diagnosed with dry socket.
2. Absence of systematic disease.

Exclusion Criteria:

1. SMOKER
2. ALCOHOLIC
3. Patients under the age of 16 years and over the age of 70 years
4. Patient with various bone diseases including osteoporosis.
5. Patients who had a history of taking oral or intravenous bisphosphonates.
6. Patients with a history of radiotherapy to the head and neck and jawbones.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 14 days
  pain will assessed using Visual Analogue scale on day 2, 6, 10 and 14th after the start of treatment. Visual Analogue Score measurement will be scale based from 1 to 10 score. Where 1-3 is mild, 3-7 is moderate and 7-10 will be scored as severe pain.
Periodontal Probe | 14 days
  alveolar osteitis affected extraction socket will be observed for the resolution of inflammation and healing will be assessed on day 2, 6, 10 and 14 by clinical examination with periodontal Probe. Periodontal depth will be measured in mm, by using the periodontal probe where the depth of 1 to 3 mm is considered well healed socket, 4-6 mm indicates moderately inflamed, 7 mm and above is considered severely inflammed .

CONTACTS AND LOCATIONS:
Overall Officials: MAIMOONA Siddiq Dr, BDS-FCPS, Study Director — Department of Oral & Maxillofacial Surgery-Dental College HITEC-IMS; Muhammad Bilal Dr, BDS, Principal Investigator — Department of Oral & Maxillofacial Surgery-Dental College HITEC-IMS
Locations (1):
- Department of Oral & Maxillofacial Surgery-Dental College HITEC-IMS TAXILA CANTT, Taxila Cantt, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
its not required for trial registry. if at any time during trial registration it is asked , i will provide the data